CLINICAL TRIAL: NCT00086476
Title: Investigations of Megakaryocytes From Patients With Abnormal Platelet Vesicles
Brief Title: Study of Megakaryocytes From Patients With Abnormal Platelet Vesicles
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040226; 04-HG-0226
Record Dates: First submitted 2004-07-01; First posted 2004-07-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-13

CONDITIONS: Blood Coagulation Disorders
Keywords: Gray Platelet Syndrome; Hermansky-Pudlak Syndrome; Storage Pool Deficiency; Organelle Formation; Megakaryocyte Development; Megakaryocytes; Platelets; Dense Granules; Alpha Granules; Lysosome-related Organelles; GPS; HPS; Griscelli Disease; Chediak Higashi Syndrome; Wiskott Aldrich Syndrome; Platelet; Congenital Bleeding Disorders; SAC; Vesicle
MeSH Terms: conditions — Blood Coagulation Disorders; Gray Platelet Syndrome; Hermanski-Pudlak Syndrome; Platelet Storage Pool Deficiency; Chediak-Higashi Syndrome; Wiskott-Aldrich Syndrome; Blister

SUMMARY:
Congenital bleeding disorders characterized by abnormal platelet granules include Gray Platelet syndrome (GPS; defective alpha-granules), Hermansky-Pudlak syndrome (HPS; defective delta-granules), and combined alpha delta-storage pool deficiency (alpha delta-SPD). Other diseases associated with variable defects in platelet gamma-granules include Chediak-Higashi, Griscelli, Wiskott-Aldrich, and Thrombocytopenia Absent Radius syndromes. These disorders are models for the study of organelle formation in megakaryocytes and platelets. Characteristics of megakaryocytopoiesis in these disorders have not been investigated because megakaryocytes could not be cultured from patients in sufficient quantities for experimental purposes. Recent advances have made it possible to culture megakaryocytes using serum-free media supplemented with recombinant human thrombopoietin (TPO). Such cultured human megakaryocytes, amplified from bone marrow-derived CD34+ stem cells, synthesize and store organellar proteins and produce functional platelets. In this protocol, we plan to obtain bone marrow aspirates from 40 children and adults (ages 2 to 80 years) with GPS, HPS, and related disorders. Patients admitted to the NIH Clinical Center on specific disease-related protocols will be enrolled in this protocol during their routine 3-5 day visits. We will culture megakaryocytes from CD34+ stem cells isolated from bone marrow aspirates. Studies of cultured megakaryocytes will include evaluation of granule membrane and soluble proteins using fluorescent antibodies and immunoelectron microscopy and comparison of RNA and protein expression patterns between normal and patient cells. Precautions will be taken to prevent the primary risk of the bone marrow aspiration, i.e., prolonged bleeding at the aspiration site. Standard diagnostic studies on the bone marrow sample may reveal information that may directly benefit patients. However, the broader benefit of this study is the acquisition of a better understanding of the characteristics of functional platelet disorders and the process of intracellular vesicle formation.

DETAILED DESCRIPTION:
Congenital bleeding disorders characterized by abnormal platelet granules include Gray Platelet syndrome (GPS; defective alpha-granules), Hermansky-Pudlak syndrome (HPS; defective delta-granules), and combined alpha delta-storage pool deficiency (alpha delta-SPD). Other diseases associated with variable defects in platelet gamma-granules include Chediak-Higashi, Griscelli, Wiskott-Aldrich, and Thrombocytopenia Absent Radius syndromes. These disorders are models for the study of organelle formation in megakaryocytes and platelets. Characteristics of megakaryocytopoiesis in these disorders have not been investigated because megakaryocytes could not be cultured from patients in sufficient quantities for experimental purposes. Recent advances have made it possible to culture megakaryocytes using serum-free media supplemented with recombinant human thrombopoietin (TPO). Such cultured human megakaryocytes, amplified from bone marrow-derived CD34+ stem cells, synthesize and store organellar proteins and produce functional platelets. In this protocol, we plan to obtain bone marrow aspirates from 40 children and adults (ages 2 to 80 years) with GPS, HPS, and related disorders. Patients admitted to the NIH Clinical Center on specific disease-related protocols will be enrolled in this protocol during their routine 3-5 day visits. We will culture megakaryocytes from CD34+ stem cells isolated from bone marrow aspirates. Studies of cultured megakaryocytes will include evaluation of granule membrane and soluble proteins using fluorescent antibodies and immunoelectron microscopy and comparison of RNA and protein expression patterns between normal and patient cells. Precautions will be taken to prevent the primary risk of the bone marrow aspiration, i.e., prolonged bleeding at the aspiration site. Standard diagnostic studies on the bone marrow sample may reveal information that may directly benefit patients. However, the broader benefit of this study is the acquisition of a better understanding of the characteristics of functional platelet disorders and the process of intracellular vesicle formation.

ELIGIBILITY:
* INCLUSION CRITERIA:

This protocol will include children and adults with a clinical diagnosis of GPS, HPS, isolated delta-SPD, combined alpha delta-SPD, Griscelli disease, Chediak Higashi syndrome, Wiskott Aldrich syndrome or Thrombocytopenia absent radius syndrome. Patients whose platelets exhibit abnormal intracellular vesicle morphology will also be eligible.

EXCLUSION CRITERIA:

Patients younger than 2 years and older than 80 years will be excluded. Patients with severe thrombocytopenia (fewer than 20 times 10(12) platelets/L) will be excluded.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-06-29; Study Completion 2011-06-13

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rendu F, Brohard-Bohn B. The platelet release reaction: granules' constituents, secretion and functions. Platelets. 2001 Aug;12(5):261-73. doi: 10.1080/09537100120068170. PMID 11487378
- [Background] White JG. Ultrastructural studies of the gray platelet syndrome. Am J Pathol. 1979 May;95(2):445-62. PMID 453324
- [Background] McNicol A, Israels SJ. Platelet dense granules: structure, function and implications for haemostasis. Thromb Res. 1999 Jul 1;95(1):1-18. doi: 10.1016/s0049-3848(99)00015-8. PMID 10403682